CLINICAL TRIAL: NCT05250349
Title: TRAnscranial Doppler CErebral Blood Flow and Cognitive IMPAIRment in Patients With Heart Failure and Presence/Absence of Atherosclerotic Carotid Artery Stenosis
Brief Title: TRAnscranial Doppler CErebral Blood Flow and Cognitive IMPAIRment in Heart Failure
Acronym: TRACE-IMPAIR
Status: Recruiting | Type: Observational
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: TRACE-IMPAIR
Record Dates: First submitted 2021-12-31; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Cognitive Impairment; Carotid Stenosis
Keywords: Carotid Stenosis; Heart Failure; Carotid Doppler; Transcranial Doppler; Cerebral Flow; Cognitive Impairment; Stroke Volume
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction; Carotid Stenosis | interventions — Echocardiography; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Isolated HF Group: Patients with echocardiography - confirmed Heart Failure (HFmrEF and HFrEF) and clinical symptoms (NYHA I-III).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Doppler sonography; Diagnostic Test: Neuropsychological tests
- HF + CS group: Patients with echocardiography - confirmed Heart Failure (HFmrEF and HFrEF) with NYHA I-III symptoms, who were diagnosed with flow limiting Carotid Stenosis on carotid Doppler ultrasound.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Doppler sonography; Diagnostic Test: Neuropsychological tests
- Control group: A cohort of patients without Heart Failure or other significant cardiac pathology and without Carotid Stenosis (a paired propensity match will be performed).
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Doppler sonography; Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Echocardiography — Transthoracic echocardiography with standard measurements
Diagnostic Test: Doppler sonography — Transcarotid and transcranial Doppler sonography
Diagnostic Test: Neuropsychological tests — Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA)

SUMMARY:
TRACE-IMPAIR is a prospective, clinical study of consecutive patients that evaluates the relationship between heart failure (HF) and cognitive impairment in relation to carotid and cerebral flow. The carotid and cerebral flow will be assessed using Doppler ultrasonography, and cognitive function will be estimated during routine neuropsychological tests.

It is an observational, three(natural)-group, single-center study. It is also an Academic Registry - the scientific activity of the Faculty of Medicine, Collegium Medicum, Jagiellonian University, and John Paul II Hospital.

DETAILED DESCRIPTION:
Circumstantial evidence suggests that cognitive dysfunction may occur in HF patients as often undiagnosed comorbidity. Cognitive dysfunction may aggravate HF symptoms and influence prognosis. Cognitive dysfunction may be a reason for inadequate self-care and poor symptom control (e.g., weight gain monitoring). In addition, it may affect medication compliance, leading to hospital readmissions and increased mortality. Brain tissue hypoxia, microemboli, silent strokes, and co-existing anemia have been implicated in contributing to cognitive dysfunction in HF. However, the role of cerebral flow impairment in these patients remains unclear. This uncertainty is mainly because previous studies included small patient groups, diverse imaging techniques, and neuropsychological tests. Furthermore, these studies were primarily conducted in the elderly, a potentially important confounder due to the effect of age on cognitive dysfunction. Particularly little data is available for younger patients (< 60 years).

This study aims to investigate the association of HF, carotid and cerebral flow, and cognitive impairment. Consecutive patients with HF with mildly reduced (HFmrEF) and reduced ejection fraction (HFrEF) will be included in the study. Echocardiography with routine measurements such as ejection fraction and stroke volume will be performed in each patient. The carotid and cerebral flow will be assessed on Doppler ultrasonography. Each patient will undergo cognitive function assessment using Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA). The results in the index group (isolated HF) will be compared with those in a group of patients with HF and flow-limiting carotid stenosis (CS) against a control group (no HF, no CS).

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients (NYHA I-III symptoms) with HF (for at least 6 months) either of ischemic or inflammatory etiology as well as genetic cardiomyopathies
* Signed informed consent form
* Consent to imaging studies: echocardiography, carotid and transcranial Doppler sonography and neuropsychological tests (MMSE and MoCA).

Exclusion Criteria:

* Co-existing, severe, irreversible disease (e.g. advanced cancer)
* Previously diagnosed dementia (including severe dementia - MMSE and MoCA score <10)
* Psychiatric condition which may influence cognitive function
* Acute, decompensated HF
* Reversible cause of HF - tachyarrhytmic, peripartum or toxic cardiomyopathy, acute myocarditis, acute myocardial infarction
* Aortic stenosis
* Cerebral stroke in the preceding 3 months
* Lack of transcranial Doppler acoustic window
* Echocardiographic projections precluding adequate measurements
* Anemia with Hemoglobin < 8 g/dl
* Alcohol or psychoactive agents abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers registry of patients with HF with mildly reduced (41-49% - HFmrEF) and reduced left ventricle ejection fraction (≤40% - HFrEF)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least moderate (i.e. mild or moderate) cognitive dysfunction (MMSE) | At six months from HF diagnosis
  Proportion of patients with at least moderate (i.e. mild or moderate) cognitive dysfunction according to Mini Mental State Examination (MMSE score ≥10)

SECONDARY OUTCOMES:
Proportion of patients with at least moderate (i.e. mild or moderate) cognitive dysfunction (MoCA) | At six months from HF diagnosis
  Proportion of patients with at least moderate (i.e. mild or moderate) cognitive dysfunction according to Montreal Cognitive Assessment (MoCA score ≥10)
Proportion of patients with mild cognitive dysfunction (MMSE) | At six months from HF diagnosis
  Proportion of patients with mild cognitive dysfunction according to Mini Mental State Examination (MMSE score 20 - 25)
Proportion of patients with mild cognitive dysfunction (MoCA) | At six months from HF diagnosis
  Proportion of patients with mild cognitive dysfunction according to Montreal Cognitive Assessment (MoCA score 18 - 25)
Proportion of patients with moderate cognitive dysfunction (MMSE) | At six months from HF diagnosis
  Proportion of patients with moderate cognitive dysfunction according to Mini Mental State Examination (MMSE score 10 - 19)4. Proportion of patients with moderate cognitive dysfunction according to Mini Mental State Examination (MMSE score 10 - 19)
Proportion of patients with moderate cognitive dysfunction (MoCA) | At six months from HF diagnosis
  Proportion of patients with moderate cognitive dysfunction according to Montreal Cognitive Assessment (MoCA score 10 - 17)
Proportion of patients with moderate reduced cerebral flow velocity | At six months from HF diagnosis
  Proportion of patients with reduced cerebral flow velocity (mean cerebral flow velocity <50 cm/s) in the middle cerebral artery among those with at least moderate (i.e. mild or moderate) cognitive dysfunction according to MMSE (MMSE score ≥10)
Proportion of patients with significantly reduced cerebral flow velocity | At six months from HF diagnosis
  Proportion of patients with reduced cerebral flow velocity (mean cerebral flow velocity <50 cm/s) in the middle cerebral artery among those with at least moderate (i.e. mild or moderate) cognitive dysfunction according to MoCA tests (MoCA score≥10)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, The John Paul II Hospital, Krakow, MP, Poland

IPD SHARING:
Plan to Share IPD: Undecided